CLINICAL TRIAL: NCT01890122
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of Alogliptin and Metformin Fixed Dose Combination, Alogliptin Alone, or Metformin Alone in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Alogliptin and Metformin Fixed-Dose Combination in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322MET_303; U1111-1139-0497 (Registry Identifier: WHO); NMRR-12-799-12754 (Registry Identifier: NMRR); CTR20130254 (Registry Identifier: SFDA CTR); 1036022140 (Registry Identifier: TCTIN)
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — alogliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metformin HCl 500 mg (Active Comparator): Metformin hydrochloride (HCl) 500 mg, capsules, orally, twice a day; alogliptin placebo-matching tablets, orally, twice a day; alogliptin and metformin HCl fixed dose combination (FDC) placebo-matching tablets, orally, twice a day for up to 26 weeks.
  Interventions: Drug: Metformin HCl; Drug: Alogliptin Placebo; Drug: Alogliptin and Metformin FDC Placebo
- Alogliptin 12.5 mg (Active Comparator): Alogliptin 12.5 mg, tablets, orally, twice a day; metformin placebo-matching capsules, orally, twice a day; alogliptin and metformin HCl FDC placebo-matching tablets, orally, twice a day for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin Placebo; Drug: Alogliptin and Metformin FDC Placebo
- Alogliptin 12.5 mg + Metformin HCl 500 mg FDC (Experimental): Alogliptin 12.5 mg and metformin HCl 500 mg FDC, tablets, orally, twice a day; alogliptin placebo-matching tablets, orally, twice a day; metformin placebo-matching capsules, orally, twice a day for up to 26 weeks.
  Interventions: Drug: Alogliptin and Metformin Fixed-Dose Combination (FDC); Drug: Alogliptin Placebo; Drug: Metformin Placebo
- Placebo (Placebo Comparator): Alogliptin and metformin FDC placebo-matching tablets, orally, twice a day; alogliptin placebo-matching tablets, orally, twice a day; metformin placebo-matching capsules, orally, twice a day for up to 26 weeks.
  Interventions: Drug: Alogliptin Placebo; Drug: Metformin Placebo; Drug: Alogliptin and Metformin FDC Placebo

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322; Nesina
  Arms: Alogliptin 12.5 mg
Drug: Metformin HCl — Metformin HCl capsules
  Other Names: Glucophage
  Arms: Metformin HCl 500 mg
Drug: Alogliptin and Metformin Fixed-Dose Combination (FDC) — Alogliptin and metformin FDC tablets
  Other Names: Kazano
  Arms: Alogliptin 12.5 mg + Metformin HCl 500 mg FDC
Drug: Alogliptin Placebo — Alogliptin placebo-matching tablets
  Arms: Alogliptin 12.5 mg + Metformin HCl 500 mg FDC; Metformin HCl 500 mg; Placebo
Drug: Metformin Placebo — Metformin placebo-matching capsules
  Arms: Alogliptin 12.5 mg; Alogliptin 12.5 mg + Metformin HCl 500 mg FDC; Placebo
Drug: Alogliptin and Metformin FDC Placebo — Alogliptin and metformin FDC placebo-matching tablets
  Arms: Alogliptin 12.5 mg; Metformin HCl 500 mg; Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of alogliptin and metformin fixed-dose combination (FDC) as compared with alogliptin alone or metformin alone on Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
The drug being tested in this study is a fixed-dose combination tablet of alogliptin and metformin to treat people who have diabetes. This study will look at glycemic control in people who take alogliptin and metformin FDC compared with alogliptin or metformin alone. The study will enroll approximately 640 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Alogliptin 12.5 mg twice daily (BID)
* Metformin hydrochloride (HCl) 500 mg BID
* Alogliptin 12.5 mg and Metformin HCl 500 mg FDC BID
* Placebo (dummy inactive pill) - this is a tablet/capsule that looks like the study drug but has no active ingredient.

All participants will be asked to take 2 tablets and 1 capsule twice a day at the same time each day throughout the study. All participants will be asked to record any hypoglycemic events in a diary. This multi-center trial will be conducted in China, South Korea, Taiwan and Malaysia. The overall time to participate in this study is 34 weeks. Participants will make 11 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a historical diagnosis of Type 2 diabetes mellitus (T2DM).
4. Male or female and aged 18 to 75 years, inclusive.
5. Body mass index (BMI) between 20 and 45 kg/m^2, inclusive.
6. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
7. Is experiencing inadequate glycemic control defined as glycosylated hemoglobin (HbA1c) concentration between 7.5% and 10%, inclusive, and has been treated with diet and exercise for at least 2 months prior to Screening. (Exception: a participant who has received any other diabetic therapy for less than 7 days in total within the 2 months prior to the screening, can be included).
8. If male, has a hemoglobin >12 g/dL (>120 g/L) at Screening or if female, has a hemoglobin >10 g/dL (>100 g/L) at Screening.
9. If male, has a serum creatinine <1.5 mg/dL at Screening or if female, has a serum creatinine <1.4 mg/dL at Screening, and estimated glomerular filtration rate (eGFR) >60 mL/min/1.73 m^2 based on calculation using the Modification of Diet in Renal Disease (MDRD) at Screening.
10. Willing and able to monitor their own blood glucose concentrations using a home glucose monitor and complete a subject diary.

Exclusion Criteria:

1. Participated in another clinical study within 90 days prior to Screening.
2. Received any investigational compound within 30 days prior to Randomization.
3. Received a dipeptidyl peptidase-4 (DPP-4) inhibitor within 3 months prior to screening.
4. History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
5. History of treatment for diabetic gastric paresis, gastric banding, or gastric bypass surgery.
6. History of diabetic ketoacidosis or hyperosmolar non-ketotic coma.
7. Chronic pancreatitis and/or history of acute pancreatitis.
8. Systolic blood pressure >180 mm Hg and/or diastolic blood pressure >110 mm Hg at Screening.
9. History of any hemoglobinopathy or diagnosis of chronic anemia.
10. New York Heart Association Class III or IV heart failure. (Participants who are stable at Class I or II and are currently treated, are candidates for the study.)
11. History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within 6 months prior to Screening.
12. History of any cancer, other than squamous cell or basal cell carcinoma of the skin, which has not been in full remission for at least 5 years prior to Screening. Participants with a history of treated cervical intraepithelial neoplasia [CIN] I or CIN II are allowed.
13. Significant clinical sign or symptom of hepatopathy, acute or chronic hepatitis, human immunodeficiency virus or alanine aminotransferase (ALT) is 2.5 times above upper limit of normal value.
14. History of angioedema in association with use of angiotensin-converting enzyme inhibitors (ACEI) or angiotensin II receptor blockers (ARB).
15. History of hypersensitivity or allergies to any DPP-4 inhibitor and/or metformin or related compounds.
16. Has used oral or systemically injected glucocorticoids (including intra-articular injection) or has used weight-loss drugs within 2 months prior to Screening. (Inhaled or topical corticosteroids were allowed.)
17. History of alcohol or substance abuse within 2 years prior to Screening.
18. Has used medicine for weight loss within 60 days prior to Screening (such as Xenical, Sibutramine, Phenylpropanolamine or similar nonprescription drugs).
19. History of organ transplantation.
20. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
21. Has, in the judgment of the investigator, any major illness or debility that may prohibit the participant from completing the study.
22. If female, is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (45):
- China (24):
  - Beijing, Beijing Municipality
  - Fuzhou, Fujian
  - Xiamen, Fujian
  - Guangzhou, Guangdong
  - Nanning, Guangxi
  - Guiyang, Guizhou
  - Hengshui, Hebei
  - Shijiazhuang, Hebei
  - Shiyan, Hubei
  - Wuhan, Hubei
  - Changsha, Hunan
  - Yueyang, Hunan
  - Changzhou, Jiangsu
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shenyang, Liaoning
  - Xi’an, Shanxi
  - Chengdu, Sichuan
  - Wenzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin
- Malaysia (12):
  - Johor Bahru, Johor
  - Alor Star, Kedah
  - Alor Star, Kedah Darul Aman
  - Kubang Kerian, Kelantan
  - Putrajaya, Kuala Lumpur
  - Kampung Baharu Nilai, Negeri Sembilan
  - Seremban, Negeri Sembilan
  - Tampin, Negeri Sembilan
  - Bagan Serai, Perak
  - Ipoh, Perak
  - Petaling Jaya, Selangor
  - Shah Alam, Selangor
- South Korea (5):
  - Goyang-si, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Busan
  - Seoul
- Taiwan (4):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei

REFERENCES:
- See also: The Alogliptin-Metformin Fixed Dose Combination (KAZANO) were approved in the United States (US) on 25 January 2013. — http://www.accessdata.fda.gov/drugsatfda_docs/label/2013/203414s000lbl.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 59 investigative sites in China, Malaysia, South Korea and Taiwan from 26 August 2013 to 05 October 2015.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes mellitus were enrolled equally in 1 of 4 treatment groups, twice a day placebo, alogliptin 12.5 mg, metformin hydrochloride (HCl) 500 mg, or alogliptin 12.5 mg and metformin HCl 500 mg fixed dose combination (FDC).
Period: Overall Study
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Started | 162 (Started = Enrolled set which included all participants who signed informed consent.) | 163 | 159 | 163
Treated | 161 (Treated = Randomized participants who received at least one dose of study drug.) | 162 | 159 | 163
Completed | 135 | 126 | 146 | 104
Not Completed | 27 | 37 | 13 | 59
Not completed — Adverse Event | 1 | 1 | 1 | 2
Not completed — Major Protocol Deviation | 3 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2
Not completed — Voluntary Withdrawal | 8 | 8 | 2 | 11
Not completed — Lack of Efficacy | 14 | 24 | 7 | 41
Not completed — Reason not Specified | 0 | 1 | 1 | 2
Not completed — Randomized but not Treated | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set consisted of all enrolled participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo | Total
Number analyzed (Participants) | 162 | 163 | 159 | 163 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.91) | 55.4 (9.62) | 53.4 (10.46) | 52.2 (10.17) | 53.6 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 65 | 68 | 68 | 281
  Male | 82 | 98 | 91 | 95 | 366
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 1 | 0 | 2 | 3
  Asian | 161 | 162 | 159 | 161 | 643
  Multiracial | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino (Yes) | 0 | 0 | 1 | 0 | 1
  Hispanic or Latino (No) | 162 | 163 | 158 | 163 | 646
Height [Mean (Standard Deviation); unit: cm] | 163.8 (8.72) | 165.0 (8.06) | 164.3 (7.66) | 164.2 (9.19) | 164.3 (8.42)
Weight [Mean (Standard Deviation); unit: kg] — Weight data is available for 161, 163, 159 and 163 participants in each treatment arm, respectively.
  kg | 70.79 (12.357) | 71.21 (11.669) | 70.73 (11.489) | 71.79 (13.949) | 71.13 (12.388)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.30 (3.566) | 26.16 (3.923) | 26.16 (3.508) | 26.56 (4.218) | 26.30 (3.811)
Smoking Classification [Number; unit: participants]
  Has Never Smoked | 125 | 112 | 113 | 112 | 462
  Is a Current Smoker | 27 | 35 | 38 | 36 | 136
  Is an Ex-smoker | 10 | 16 | 8 | 15 | 49
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 47 | 45 | 37 | 45 | 174
  Surgically Sterile | 8 | 8 | 10 | 5 | 31
  Female of Childbearing Potential | 25 | 12 | 21 | 18 | 76
  Not Applicable (Participant is Male) | 82 | 98 | 91 | 95 | 366
Region of Enrollment [Number; unit: participants]
  China | 129 | 129 | 128 | 130 | 516
  Korea, Republic of | 9 | 10 | 10 | 10 | 39
  Malaysia | 19 | 19 | 18 | 19 | 75
  Taiwan, Province of China | 5 | 5 | 3 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26 (or Early Termination)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 26 or early termination relative to baseline. Negative change indicates better glycemic control.
Time Frame: Baseline and Week 26 (or Early termination)
Population: Full analysis set consisted of all randomized participants in the safety set (participants who received at least 1 dose of study drug) who had baseline and at least 1 post baseline assessment. Last observation carried forward (LOCF) imputation was utilized.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 160 | 160 | 158 | 157
percentage of glycosylated hemoglobin | -0.32 (1.067) | -1.23 (0.877) | -1.06 (0.970) | -1.72 (1.024)
Statistical Analysis 1: Comparison: Metformin HCl 500 mg vs Alogliptin 12.5 mg + Metformin HCl 500 mg FDC; Test type: Superiority or Other; p < 0.0001, ANCOVA — An analysis of covariance (ANCOVA) model was used with treatment and country as fixed effects, and Baseline HbA1c as a continuous covariate; Least Square Mean Difference = -0.49, 95% CI 2-sided [-0.700 to -0.278], Standard Error of Mean 0.107
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg vs Alogliptin 12.5 mg + Metformin HCl 500 mg FDC; Test type: Superiority or Other; p < 0.0001, ANCOVA — An ANCOVA model was used with treatment and country as fixed effects, and Baseline HbA1c as a continuous covariate; Least Square Mean Difference = -0.68, 95% CI 2-sided [-0.889 to -0.467], Standard Error of Mean 0.108

2. Secondary Outcome: Change From Baseline in HbA1c at Weeks 4, 8, 12, 16 and 20
Description: The change in the value of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Weeks 4, 8, 12, 16 and 20 relative to baseline. Negative change indicates better glycemic control.
Time Frame: Baseline and Weeks 4, 8, 12, 16 and 20
Population: Full analysis set consisted of all randomized participants in the safety set (participants who received at least 1 dose of study drug) who had baseline and at least 1 post baseline assessment. LOCF imputation was utilized. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of glycosylated hemoglobin
  Week 4 (n=157,156,154,156) | -0.57 (0.483) | -0.41 (0.570) | -0.80 (0.489) | -0.18 (0.503)
  Week 8 (n=160,160,158,157) | -0.90 (0.682) | -0.78 (0.756) | -1.29 (0.732) | -0.29 (0.738)
  Week 12 (n=160,160,158,157) | -1.06 (0.793) | -1.01 (0.839) | -1.57 (0.873) | -0.27 (0.895)
  Week 16 (n=160,160,158,157) | -1.18 (0.816) | -1.06 (0.900) | -1.71 (0.937) | -0.33 (0.957)
  Week 20 (n=160.160,158,157) | -1.24 (0.852) | -1.11 (0.925) | -1.74 (0.969) | -0.33 (1.006)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 4, 8, 12, 16, 20 and 26
Description: The change between the FPG value collected at Weeks 4, 8, 12, 16, 20 and 26 relative to baseline. Negative change indicates better glycemic control.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
mg/dL
  Week 4 (n=157,154,155,156) | -1.42 (1.344) | -1.01 (1.794) | -2.01 (2.157) | 0.02 (1.532)
  Week 8 (n=160,158,158,157) | -1.50 (1.571) | -1.17 (1.788) | -2.13 (1.808) | -0.08 (1.682)
  Week 12 (n=160,158,158,157) | -1.48 (1.527) | -1.33 (1.938) | -2.14 (1.779) | -0.08 (2.112)
  Week 16 (n=160,158,158,157) | -1.62 (1.599) | -1.25 (2.148) | -2.17 (1.923) | -0.07 (2.020)
  Week 20 (n=160,158,158,157) | -1.57 (1.634) | -1.19 (2.248) | -2.26 (1.995) | -0.12 (2.092)
  Week 26 (n=160,158,158,157) | -1.45 (1.674) | -1.06 (2.307) | -2.06 (2.274) | -0.04 (2.060)

4. Secondary Outcome: Time to Hyperglycemic Rescue Event
Description: Rescue is defined as meeting one of the following criteria, confirmed by a second sample drawn within 7 days of first sample: After >1 week of treatment but prior to Week 4 visit: A single FPG ≥275 mg/dL (≥15.27 mmol/L); From the Week 4 but prior to the Week 8 visit: A single FPG ≥250 mg/dL (≥13.88 mmol/L); From the Week 8 visit but prior to the Week 12 visit: A single FPG ≥225 mg/dL (≥12.49 mmol/L); From the Week 12 visit through the end-of-treatment visit (week 26): HbA1c ≥8.5% and ≤0.5% reduction in HbA1c from baseline. Time to hyperglycemic rescue was censored if the participant did not experience a hyperglycemic rescue event.
Time Frame: From the date of randomization through Week 26
Population: Randomized set consisted of all enrolled participants who were randomized.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 162 | 162 | 159 | 163
days | NA [NA to NA] — Data was not estimable as fewer than 50% of participants in any arm required hyperglycemic rescue. | NA [NA to NA] — Data was not estimable as fewer than 50% of participants in any arm required hyperglycemic rescue. | NA [NA to NA] — Data was not estimable as fewer than 50% of participants in any arm required hyperglycemic rescue. | NA [113.0 to NA] — Data was not estimable as fewer than 50% of participants in any arm required hyperglycemic rescue.

5. Secondary Outcome: Percentage of Participants Requiring Hyperglycemic Rescue
Description: Rescue is defined as meeting one of the following criteria, confirmed by a second sample drawn within 7 days of first sample: After >1 week of treatment but prior to Week 4 visit: A single FPG ≥275 mg/dL (≥15.27 mmol/L); From the Week 4 but prior to the Week 8 visit: A single FPG ≥250 mg/dL (≥13.88 mmol/L); From the Week 8 visit but prior to the Week 12 visit: A single FPG ≥225 mg/dL (≥12.49 mmol/L); From the Week 12 visit through the end-of-treatment visit (week 26): HbA1c ≥8.5% and ≤0.5% reduction in HbA1c from baseline.
Time Frame: Baseline up to Week 26
Population: Full analysis set consisted of all randomized participants in the safety set (participants who received at least 1 dose of study drug) who had baseline and at least 1 post baseline assessment. LOCF imputation was utilized.
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 8.7 | 14.8 | 4.4 | 25.5

6. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia
Description: Marked hyperglycemia is defined as FPG level ≥200 mg/dL (11.1 mmol/L).
Time Frame: Baseline up to Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 8.8 | 12.7 | 5.7 | 15.9

7. Secondary Outcome: Change From Baseline in Body Weight at Weeks 12 and 26
Description: Change in participant's body weight at Weeks 12 and 26 relative to baseline.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: kg
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 158
kg
  Week 12 (n=153,151,149,145) | -0.71 (1.735) | -0.19 (1.696) | -0.14 (1.730) | -0.32 (1.837)
  Week 26 (n=156,156,156,152) | -0.93 (2.240) | -0.22 (2.291) | -0.57 (2.336) | -0.33 (2.220)

8. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤6.5%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) ≤6.5%.
Time Frame: Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 27.3 | 21.6 | 55.1 | 11.8

9. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤7.0%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) ≤7%.
Time Frame: Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 55.9 | 44.4 | 77.2 | 30.4

10. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤7.5%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) ≤7.5%.
Time Frame: Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 73.3 | 60.5 | 84.8 | 46.0

11. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥0.5%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with a decrease from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) of ≥0.5%.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 81.4 | 74.1 | 89.2 | 42.9

12. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥1.0%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with a decrease from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) of ≥1.0%.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 63.4 | 53.7 | 83.5 | 25.5

13. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥1.5%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with a decrease from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) of ≥1.5%.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 37.3 | 36.4 | 62.0 | 14.9

14. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥2.0%
Description: Clinical response at Week 26 will be assessed by the percentage of participants with a decrease from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) of ≥2.0%.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Number analyzed (Participants) | 161 | 162 | 158 | 161
percentage of participants | 17.4 | 17.3 | 34.8 | 6.2

ADVERSE EVENTS:
Time Frame: Week 1 up to Week 28
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety set, all participants who took at least 1 dose of double-blind study drug.
Arm/Group | Metformin HCl 500 mg | Alogliptin 12.5 mg | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC | Placebo
Serious Adverse Events (participants affected / at risk) | 5/161 | 4/162 | 4/158 | 5/161
Other Adverse Events (participants affected / at risk) | 33/161 | 26/162 | 25/158 | 35/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin HCl 500 mg (N=161) | Alogliptin 12.5 mg (N=162) | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC (N=158) | Placebo (N=161)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with placebo and is not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin HCl 500 mg (N=161) | Alogliptin 12.5 mg (N=162) | Alogliptin 12.5 mg + Metformin HCl 500 mg FDC (N=158) | Placebo (N=161)
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 11 | 8 | 8 | 9
Nasopharyngitis (Infections and infestations) | 6 | 3 | 2 | 6
Protein urine present (Investigations) | 5 | 2 | 7 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 9 | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.